CLINICAL TRIAL: NCT03610256
Title: Prospective Multicentric Randomized Trial Comparing the Efficacy and Safety of Single-anastomosis Duodeno Ileal Bypass With Sleeve Gastrectomy (SADI-S) Versus Roux-en-Y Gastric Bypass (RYGB)
Brief Title: Single-anastomosis Duodeno Ileal Bypass (SADI) Versus Roux-en-Y Gastric Bypass
Acronym: SADISLEEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0042; 2018-A01051-54 (Other: ID-RCB)
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Bariatric surgery; Single-anastomosis duodeno ileal bypass (SADI); Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SADI-S (Experimental): This corresponds to obese patients (BMI ≥40 kg/m2 or BMI ≥35 kg/m2 +/- co-morbidities (high blood pressure, dyslipidemia, obstructive sleep apnea, type 2 diabetes mellitus, arthrosis)) benefiting from a laparoscopic SADI-S (laparoscopic Single-anastomosis duodeno ileal bypass with Sleeve gastrectomy).
  SADI-S will be performed as a primary procedure or after failure of sleeve gastrectomy, defined as insufficient weight loss at 18 months after surgery (EWL% <50), or as weight regain (+ 20% of nadir weight).
  Interventions: Procedure: SADI-S
- RYGB (Active Comparator): This corresponds to obese patients (BMI ≥40 kg/m2 or BMI ≥35 kg/m2 +/- co-morbidities (high blood pressure, dyslipidemia, obstructive sleep apnea, type 2 diabetes mellitus, arthrosis)) benefiting from a laparoscopic RYGB (laparoscopic Roux-en-Y Gastric ByPass).
  Similarly to the experimental group, RYGB will be performed as a primary procedure or after failure of sleeve gastrectomy, which is defined as insufficient weight loss at 18 months after surgery (EWL% <50), or as weight regain (+ 20% of nadir weight).
  Interventions: Procedure: RYGB

INTERVENTIONS:
Procedure: SADI-S — Laparoscopic SADI-S, recently described as an evolution of the BPD-DS, combining the physiological advantages of pylorus preservation and the technical benefits of single-loop reconstruction, associating a sleeve gastrectomy and a duodeno-ileal bypass at 2.5 meters from the ileo-caecal valve if BMI ≥ 50 kg/m² or at 3 meters if BMI < 50
  Other Names: Laparoscopic Single-anastomosis duodeno ileal bypass with Sleeve gastrectomy (SADI-S)
  Arms: SADI-S
Procedure: RYGB — The laparoscopic Roux-en-Y Gastric Bypass will consist of:
  * a small gastric pouch (about 30cc)
  * an antecolic alimentary limb
  * a gastro-jejunal anastomosis using a linear stapler
  * a 150cm long alimentary limb
  * a 50cm biliary limb
  * a latero-lateral jejuno-jejunal anastomosis
  * closure of the mesenteric defects
  Other Names: Roux-en-Y Gastric ByPass
  Arms: RYGB

SUMMARY:
Obesity is a major public health problem worldwide. Bariatric surgery has proved to be the most effective treatment of morbid obesity in terms of weight reduction and remission of co-morbid conditions during long-term follow-up. Nowadays, France is ranked 3rd in terms of bariatric surgeries performed per year.

Since the laparoscopic Roux-en-Y gastric bypass (RYGB) was described in 1977, this restrictive and malabsorptive procedure has become a gold standard for morbid obesity with an average Excess Weight Loss % (EWL%) of 72% at 2 years, and a strong metabolic effect, especially with regard to type 2 diabetes remission. Nevertheless, failures are observed (up to 20%), particularly in super obese patients, which are then difficult to manage. In this population, biliopancreatic diversion with duodenal switch (BPD-DS) is indicated due to its stronger weight loss and metabolic effect, but is still little performed worldwide because of its higher morbidity, surgical complexity and risk of malnutrition.

A novel technique combining the physiological advantages of pylorus preservation and the technical benefits of single-loop reconstruction was introduced in 2007 by Sanchez-Pernaute, who described the single-anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S) as an evolution of the BPD-DS. With a 2.5-meter common channel, SADI-S seems to offer good results for the treatment of both morbid obesity and its metabolic complications, with an EWL% of up to 95% at 2 years and potentially less nutritional consequences.

To date, there is only one Spanish randomized trial comparing SADI-S to BPD-DS, whereas BPD-DS represents less than 1% of bariatric procedures in France and is only allowed in super obese patients. Thus only preliminary data of poor scientific value exists. Nevertheless, facing very encouraging short-term outcomes, there is a real need for a prospective trial comparing SADI-S to a standard bariatric procedure.

The aim of the investigator's study is to assess weight loss efficiency and the morbi-mortality of the SADI-S in comparison to a standard (RYGB), in order to validate this procedure among bariatric techniques

HYPOTHESIS SADI-S is superior to the standard RYGB for weight loss, increasing the EWL% by 10% (82% vs 72%, respectively) at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 65 years old,
* Morbid obesity with BMI ≥40 kg/m2 or BMI ≥35 kg/m2 associated with one co-morbidity which will be improved by surgery (high blood pressure, type 2 diabetes mellitus, obstructive sleep apnea, dyslipidemia, arthrosis)
* Patient who has benefited from an upper GI endoscopy with biopsies to look for Helicobacter pylori , within the 12 months before surgery,
* Patient who has benefited from a pluridisciplinary evaluation, with a favorable opinion for SADI-S or RYGB as a primary surgery or after failure of sleeve gastrectomy (defined as insufficient weight loss at 18 months after surgery (EWL% <50), or as weight regain (+ 20%)).
* Patient who understands and accepts the need for a long term follow-up,
* Patient who agrees to be included in the study and who signs the informed consent form,
* Patient affiliated with a healthcare insurance plan.

Exclusion Criteria:

* History of previous bariatric surgery, other than a sleeve gastrectomy,
* Presence of a severe and evolutive life threatening pathology, unrelated to obesity,
* History of type 1 diabete,
* History of chronic inflammatory bowel disease,
* Pregnancy or desire to be pregnant during the study,
* Presence of Helicobacter pylori resistant to medical treatment,
* Presence of a unhealed gastro-duodenal ulcer or diagnosed less than 2 months previously,
* Mentally unbalanced patients, under supervision or guardianship,
* Patient who does not understand French/ is unable to give consent,
* Patient not affiliated to a French or European healthcare insurance,
* Patient who has already been included in a trial which has a conflict of interests with the present study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Excess Weight Loss measurement | 2 years after surgery
  For each surgical procedure, weight loss will be assessed 2 years after surgery using Excess Weight Loss percentage (EWL%), calculated using the following formula:
  ((weight at 2-year visit - initial weight) / (initial weight - ideal weight)) X 100 The assessment of the primary endpoint will be standardized between the centers and carried out under blind conditions.

SECONDARY OUTCOMES:
Albumin | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of albumin will explore the nutritional status of patients. Results will be expressed in g/l
Pre-albumin | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of pre-albumin will explore the nutritional status of patients. Results will be expressed in g/l
Hemoglobin | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of Hemoglobin will explore the nutritional status of patients. Results will be expressed in g/l
Calcium | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of Calcium will explore the nutritional status of patients. Results will be expressed in mmol/l
Ferritin | At each study visit (before surgey and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of ferritin will explore the nutritional status of patients. Results will be expressed in microg/l
Iron | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of iron will explore the nutritional status of patients. Results will be expressed in micromol/l
% of transferrin saturation | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of % of transferrin saturation will explore the nutritional status of patients. Results will be expressed in %
Vitamin A | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of vitamin A will explore the nutritional status of patients. Results will be expressed in micromol/l
Vitamin B1 | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of vitamin B1 will explore the nutritional status of patients. Results will be expressed in nmol/l
Vitamin B12 | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of vitamin B12 will explore the nutritional status of patients. Results will be expressed in pmol/l
Vitamin B9 | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of vitamin B9 will explore the nutritional status of patients. Results will be expressed in nmol/l
Vitamin D | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of vitamin D will explore the nutritional status of patients. Results will be expressed in nmol/l
Vitamin C | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of vitamin C will explore the nutritional status of patients. Results will be expressed in micromol/l
Vitamin E | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of vitamin E will explore the nutritional status of patients. Results will be expressed in micromol/l
Prothrombin rate | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Measurement of prothrombine rate will explore the nutritional status of patients. Results will be expressed in %
Steatorrhea rate | 6 month after surgery
  Measurement of the 24-hour steatorrhea rate will explore the nutritional status of patients. Results will be expressed in grams of lipids /100g of stools
Average number of stools per day | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of the average number of stool will explore the nutritional status of patients. Results will be expressed in number of stool/day
HbA1c | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of HbA1c will explore the Metabolic efficiency of surgery. Results will be expressed in %
Fasting glycemia | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of fasting glycemia will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
HDL | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of HDL will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
LDL | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of LDL will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
Cholesterol | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of cholesterol will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
Triglycerides | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Measurement of triglycerides will explore the Metabolic of surgery. Results will be expressed in mmol/l
Antidiabetic drugs | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Evolution of antidiabetic drugs will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Antilipidemic drugs | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Evolution of antilipidemic drugs will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Antihypertensive drugs | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Evolution of antihypertensive drugs will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Use of Continuous Positive Airway Pressure for Obstructive Sleep Apnea | Before surgery and 6, 12, 24, 60 and 120 months after surgery
  Evolution of the use of Continuous Positive Airway Pressure for Obstructive Sleep Apnea will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of persistence or not of obstructive sleep apnea.
Length of stay | End of the hospitalization period
  The Length of stay (in days) is based on the number of days of hospitalization from surgery (day of surgery = D0) until the end of hospitalization.
Readmission of patient | 30 days after surgery
  Number of patients readmitted within 30 days after surgery.
Occurrence of kidney stones | Within 10 years after surgery
  For each visit after the surgery, the presence or not of kidney stones will be documented and if applicable the treatment will be noted
Overall complication rate | Within 10 years after surgery
  Rate of medical and surgical (> or = grade 3) complications within 120 months after surgery using the Dindo-Clavien classification, described as :
  Grade I = Any deviation from the normal postoperative course. Grade 2 = Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III = Requiring surgical, endoscopic or radiological intervention, not under (Grade IIIa) or under general anesthesia (Grade IIIb) Grade IV = Life-threatening complication with single organ (Grade IVa) or Multiorgan dysfunction (Grade IVb) Grade V = Death of a patient.
Type and severity of early complications | Within 30 days after surgery
  Type (medical or surgical) and severity of early complications (within 30 days) for each procedure according to the Dindo-Clavien classification (description of this classification was made in outcome 32).
Type and severity of late complications | Within 10 years after surgery
  Type (medical or surgical) and severity of late complications (after 30 days) for each procedure according to the Dindo-Clavien classification (description of this classification was made in outcome 32).
Gastroesophageal reflux assessment | At each study visit (before surgery and 1, 3, 6, 12,18, 24, 60 and 120 months after surgery)
  Evolution of gastroesophageal reflux will be assessed at each study visit, before and after surgery. This outcome will be expressed in terms of improvement, aggravation or onset.
Absolute weight loss assessment | 1, 3, 6, 12, 18, 24, 60 and 120 months after surgery
  Weight loss at 1, 3, 6, 12, 18, 24, 60 and 120 months after surgery, according to absolute weight loss (aWL) in kg.
Excess Weight Loss percentage assessment | 1, 3, 6, 12, 18, 24, 60 and 120 months after surgery
  Weight loss at 1, 3, 6, 12, 18, 24, 60 and 120 months after surgery, according to Excess Weight Loss percentage (EWL%), calculated using the following formula:
  ((weight at visit X - initial weight) / (initial weight - ideal weight)) X 100
Excess BMI Loss percentage assessment | 1, 3, 6, 12, 18, 24, 60 and 120 months after surgery
  Weight loss at 1, 3, 6, 12, 18, 24, 60 and 120 months after surgery, according Excess BMI Loss percentage (EBL%), according to the formula :
  ((BMI at visit X - initial BMI) / (initial BMI - ideal BMI)) X 100 with Ideal BMI = 25 kg/m²
Quality of life assessed with GIQLI questionnaire | Before surgery and at 6, 12 and 24 months after surgery
  Before surgery and at 6, 12 and 24 months after surgery, according to the GIQLI questionnaire.
  This questionnaire consists of 36 items exploring 5 dimensions or subscales: symptoms, physical condition, emotions, social integration and the effect of any medical treatment. For each item, 5 responses will be proposed to the patients and for each answer, a score ranging from 0 to 4 (highest score = 144) will be assigned. A high score defines a more favorable health state.
Quality of life assessed with SF36 questionnaire | Before surgery and at 6, 12 and 24 months after surgery
  Before surgery and at 6, 12 and 24 months after surgery, according to the SF36 questionnaire.
  This questionnaire taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/tiredness, and general health perceptions. It also includes a single item that provides an indication of a perceived change in health
Quality of life assessed with Sigstad questionnaire | Before surgery and at 1, 3, 6, 12, 24, 60 and 120 months after surgery
  Sigstad questionnaire for all postoperative study visits (except 18 months after surgery).
  The Sigstad questionnaire allows the identification and diagnosis of postoperative dumping syndrome and early hypoglycaemia: a score >7 suggests a dumping syndrome
Evolution of food choices and preferences within 2 years after surgery | Before surgery and 3, 12 and 24 months after surgery
  The evolution of food choices and preferences will be measured before surgery and 3, 12 and 24 months after surgery using a computerized test: the "Leeds Food Preference Questionnaire (LFPQ).
  The Leed Food Preference Questionnaire provides measurements of different components of food preference and food reward, and is a computerized questionnaire. Participants are presented with an array of pictures of individual food items common in the diet. Foods are chosen from a validated database to be either predominantly high (>50% energy) or low (<20% energy) in fat but similar in familiarity, protein content, sweet or not-sweet taste and palatability. Responses are recorded and used to compute mean scores for high fat, low fat, sweet or savory food types (and different fat-taste combinations).
  This assessment will be performed only in the coordinating center
Modifications of the gastric and esophageal mucosa | 60 and 120 months after surgery
  Macroscopic data and Histological modifications of the gastric and esophageal mucosa based on upper GI endoscopy with biopsies of the gastric and esophageal mucosa
Number of reflux episodes | 60 and 120 months after surgery
  Number of reflux episodes for assessment of severe GastroEsophageal Reflux Disease by pHmetry
Number of reflux episodes lasting more than 5 minutes | 60 and 120 months after surgery
  Number of reflux episodes lasting more than 5 minutes for assessment of severe GastroEsophageal Reflux Disease by pHmetry
Exposure time with pH < 4 | 60 and 120 months after surgery
  % of exposure time with pH < 4 for assessment of severe GastroEsophageal Reflux Disease by pHmetry
Number of acid refluxes | 60 and 120 months after surgery
  Number of acid refluxes for assessment of severe GastroEsophageal Reflux Disease by pH- impedancemetry
Number of non-acid refluxes | 60 and 120 months after surgery
  Number of non-acid refluxes for assessment of severe GastroEsophageal Reflux Disease by pH- impedancemetry
Number of poor acid reflux | 60 and 120 months after surgery
  Number of poor acid reflux for assessment of severe GastroEsophageal Reflux Disease by pH- impedancemetry
Association with symptoms | 60 and 120 months after surgery
  Positive association with symptoms for assessment of severe GastroEsophageal Reflux Disease by pH- impedancemetry

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - Département de Chirurgie Digestive et Viscérale - Clinique de l'Anjou, Angers
  - Service de Chirurgie Digestive et Endocrinienne - Groupe Hospitalier Pellegrin, Bordeaux
  - Service de Chirurgie Digestive et Viscérale - Clinique La Parisière, Bourg-de-Péage
  - Département de Chirurgie Digestive et Viscérale, Centre Hospitalier Jean Marcel, Brignoles
  - Département de Chirurgie Digestive, Centre Hospitalier René Dubos, Cergy-Pontoise
  - Département de Chirurgie Digestive et Thoracique, Hôpitaux Civils de Colmar, Colmar
  - Service de Chirurgie Générale et Digestive - Hôpital Louis Mourier, Colombes
  - Service de Chirurgie Digestive - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Département de Chirurgie Digestive - CHU Grenoble, Grenoble
  - Service de Chirurgie Générale et Endocrinienne - Hôpital Huriez, Lille
  - Service de Chirurgie Digestive et Bariatrique - Hôpital Edouard Herriot - HCL, Lyon
  - Service de Chirurgie Digestive et Endocrinienne - Hôtel Dieu, Nantes
  - Service de Chirurgie Digestive et Transplantation - Hôpital Archet II, Nice
  - Département de Chirurgie Digestive et Hépatobiliaire - Hôpital Pitié Salpétrière, Paris
  - Département de Chirurgie Digestive - Institut Mutualiste Montsouris, Paris
  - Service de Chirurgie Digestive - Hôpital Bichat, Paris
  - Service de Chirurgie Digestive, Générale et Cancérologique - HEGP, Paris
  - Service d'Endocrinologie, Diabète et Nutrition - Centre Hospitalier Lyon Sud - HCL, Pierre-Bénite
  - Département de Chirurgie Digestive et Hépatobiliaire - Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire
  - Département de Chirurgie Digestive et Bariatrique, Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Service de Chirurgie Digestive, Hôpital Rangueil, Toulouse
  - Service de Chirurgie Digestive, Hépatobiliaire et Endocrinienne - Hôpital Brabois adultes, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Robert M, Poghosyan T, Delaunay D, Pelascini E, Iceta S, Sterkers A, Barsamian C, Khamphommala L, Bin Dorel S, Maucort-Boulch D, Czernichow S, Disse E. Prospective multicentre randomised trial comparing the efficacy and safety of single-anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S) versus Roux-en-Y gastric bypass (RYGB): SADISLEEVE study protocol. BMJ Open. 2020 Sep 1;10(9):e037576. doi: 10.1136/bmjopen-2020-037576. PMID 32873678
- [Result] Robert M, Poghosyan T, Romain-Scelle N, Czernichow S, Delaunay D, Sterkers A, Khamphommala L, Lazzati A, Blanchard C, Caiazzo R, Pattou F, Disse E; SADISLEEVE Collaborative Group. Efficacy and safety of single-anastomosis duodeno-ileal bypass with sleeve gastrectomy versus Roux-en-Y gastric bypass in France (SADISLEEVE): results of a randomised, open-label, superiority trial at 2 years of follow-up. Lancet. 2025 Aug 23;406(10505):846-859. doi: 10.1016/S0140-6736(25)01070-0. PMID 40849141
- [Derived] Osorio J, Lazzara C, Guimaraes M, Torres A, Turrado-Rodriguez V, Ibarzabal A, Sobrino L, Nora M, Vilarrassa N, de Hollanda A, Rubio-Herrera MA, Vidal J, Moize V, Yarnoz C, Fernandez-Falop I, Portillo M, Sanchez-Pernaute A. A randomized open-label multicentre clinical trial comparing single-anastomosis duodenal switch (SADI-S) versus Roux-en-Y gastric bypass for the treatment of severe obesity: BYPSADIS study protocol. Scand J Surg. 2025 Oct 17:14574969251385873. doi: 10.1177/14574969251385873. Online ahead of print. PMID 41104829